CLINICAL TRIAL: NCT02679235
Title: Brain Energy and Aging With Triheptanoin: The BEAT7 Study
Brief Title: Brain Energy and Aging With Triheptanoin
Acronym: BEAT7
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-617; 188505 (Registry Identifier: Office of Clinical Trials - Health Canada)
Record Dates: First submitted 2016-02-01; First posted 2016-02-10 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Frontal Lobe Hypometabolism

STUDY DESIGN:
Intervention Model Description: The participant will receive THN treatment, compared to PRE supplementation condition.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triheptanoin (Experimental): Participant will undergo POST Triheptanoin suppementation 1g/kg body weight for 28 days (dose gradually increased each week, starting at, 0.25, 0.5, 0.75 and then 1 g) separated in 4 doses (with eah meal and before night) after a control PRE supplementation imaging protocol.
  Interventions: Drug: POST Triheptanoin

INTERVENTIONS:
Drug: POST Triheptanoin — The target daily dose of triheptanoin will be 1 g/kg/d, or approximately 70 g/d during 28±2 days. It will be divided into four daily doses, one of which will be consumed at each meal and one with an evening snack.
  Other Names: POST THN

SUMMARY:
BEAT7-001 is a single group study (supplementation). Using a multi-modal brain imaging portfolio, this study will assess whether brain energy metabolism (glucose and ketones), structure or functional connectivity change in older people with frontal glucose hypometabolism after 28 days on an oral dose of 1 g/kg/day of triheptanoin.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥65 years old;
* Score ≥26/30 on the Montreal Cognitive Assessment; -≥10% lower brain glucose uptake in the frontal cortex as determined by PET imaging.

Exclusion Criteria:

* Score <26/30 on the Montreal Cognitive Assessment;
* Medications likely to affect the primary cognitive outcome;
* Medical or psychiatric conditions that could interfere with study participation (Peterson et al. 2005);
* Fasting plasma glucose ≥7.0 mM (to avoid recruiting diabetics or pre-diabetics, both of which are risk factors for cognitive impairment in older persons (Mortimer et al. 2010) and also inhibit ketogenesis (Fukao et al. 2004);
* Clinically-significant gastro-intestinal disease/conditions;
* Clinically-significant liver disease/dysfunction : ALT ≥37 UI/L, AST ≥36 UI/L, Total bilirubin ≥26 μmol/L;
* Clinically-significant renal disease/dysfunction : creatinine ≥92 μmol/L, glomerular filtration rate <60 ml/min/1.73 m2 or >90 ml/min/1.73 m2;
* Clinically-significant cardiac disease/conditions;
* Clinically-significant abnormal coagulation laboratory results or coagulation disorders at screening;
* Poorly controlled dyslipidemia (total cholesterol ≥6.2 mmol/L or triglycerides ≥2.20 mmol/L)
* Hypertension: ≥140/90 mmHg;
* Substance abuse;
* Already on MCT supplementation;
* Visual or hearing impairment impeding comprehension;
* Non-French speaking;
* Any condition with life expectancy less than 5 years;
* Institutionalized or intending to move out of area within 1 year;
* Participation in other intervention trials.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, Ph.D., Principal Investigator — Research Centre on Aging (CSSS-IUGS - CIUSSS de l'Estrie - CHUS)
Locations (1):
- Research Centre on Aging (CSSS-IUGS - CIUSSS de l'Estrie - CHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Triheptanoin: Participant will undergo POST Triheptanoin suppementation 1g/kg body weight for 28 days (dose gradually increased each week, starting at, 0.25, 0.5, 0.75 and then 1 g) separated in 4 doses (with eah meal and before night) after a control PRE supplementation imaging protocol.
  POST Triheptanoin: The target daily dose of triheptanoin will be 1 g/kg/d, or approximately 70 g/d during 28±2 days. It will be divided into four daily doses, one of which will be consumed at each meal and one with an evening snack.
  control PRE supplementation: Before supplementation, same participants will undergo imaging protocol as a control condition. Participant will be asked to follow daily normal routine, without any change in medication or food habit.
Period: Overall Study
Arm/Group | Triheptanoin
Started | 15
Completed | 11
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Only the 11 participants which have completed the intervention are included in the baseline analysis
Arm/Group | Triheptanoin
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Glucose uptake changes estimated by comparing participants' measurements to imaging standards of hea [Mean (Standard Deviation); unit: % of difference compare to young control] | -14.8 (3.9)
Education [Mean (Standard Deviation); unit: years] | 16.5 (3.0)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: scores on a scale] — Assessment of cognition. The scale ranges from 0 to 30 points, with higher scores representing better cognitive ability
  scores on a scale | 27.3 (2.6)
body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Global Change in Brain Glucose Uptake
Description: Global change (average of cortex) in brain glucose uptake as measured by 18F-FDG PET scans PRE vs POST 28±2 days of supplementation
Time Frame: 28±2 days
Measure: Mean (Standard Deviation); unit: μmol/100 g/min
Arm/Group | Triheptanoin
Number analyzed (Participants) | 11
μmol/100 g/min
  PRE | 30.3 (1.7)
  POST supplementation | 30.4 (3.4)

2. Primary Outcome: Global Change in Brain Ketone Uptake
Description: Global change in brain ketone uptake as measured by 11C-acetoacetate PET scans
Time Frame: 28±2 days
Measure: Mean (Standard Deviation); unit: μmol/100 g/min
Arm/Group | Triheptanoin
Number analyzed (Participants) | 11
μmol/100 g/min
  PRE | 0.58 (0.4)
  POST supplementation | 0.26 (0.2)

3. Secondary Outcome: Change in Brain Volumes
Description: Structural imaging by T1-weighted MRI to measure brain volume
Time Frame: 28±2 days
Population: data was not available for 2 participants
Measure: Mean (Standard Deviation); unit: ml/100 g/ min
Arm/Group | Triheptanoin
Number analyzed (Participants) | 9
ml/100 g/ min
  hipocampus PRE | 7.4 (0.7)
  hipocampus POST supplementation | 7.4 (0.7)
  Amygdala PRE | 3.0 (0.5)
  Amygdala POST supplementation | 3.0 (0.5)
  Thalamus PRE | 12.8 (1.3)
  Thalamus POST suplementation | 12.5 (1.2)
  Caudate PRE | 6.9 (0.8)
  Caudate POST supplementation | 6.8 (0.7)

4. Secondary Outcome: Change in Cerebral Blood Flow
Description: change in cerebral blood flow measured by arterial spin labeling (ASL) and calculated using a one-compartment model (average cortex)
Time Frame: 28±2 days
Measure: Mean (Standard Deviation); unit: ml/100 g/ min
Arm/Group | Triheptanoin
Number analyzed (Participants) | 11
ml/100 g/ min
  PRE | 41.8 (9.1)
  POST supplementation | 41.8 (9.4)

ADVERSE EVENTS:
Time Frame: During 4 week supplementation period
Arm/Group | Triheptanoin
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triheptanoin (N=15)
severe stomach pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT02679235/Prot_SAP_000.pdf